CLINICAL TRIAL: NCT07353879
Title: Exploring the Effects of a Computerized Naming Intervention Combined With Cerebellar tDCS in Cantonese-Speaking Individuals With Aphasia
Brief Title: Application of Cerebellar tDCS in Aphasia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Hong Kong (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: EAU23035
Record Dates: First submitted 2025-12-29; First posted 2026-01-21 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2023-12

CONDITIONS: Aphasia Following Cerebral Infarction
Keywords: Aphasia; Non-Invasive Brain Stimulation; Transcranial Direct Current Stimulation; Cerebellum; Stroke Rehabilitation; Computerized intervention; Speech Perception training; Naming intervention; Noun naming; Verb naming
MeSH Terms: conditions — Aphasia

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active tDCS (Experimental): Cerebellar tDCS is delivered using a Soterix Medical MxN High Definition tDCS Stimulator. Real tDCS is applied to the right posterolateral cerebellum, with one anodal electrode (2 mA) placed at PO10 and two return electrodes (-1 mA each) at P10 and O10, using EEG-sized electrodes (external diameter of 1.2 cm) secured in an EEG cap. For real tDCS, participants receive five sessions, each consisting of 20 minutes of 2 mA anodal stimulation with 30-second ramp-up and ramp-down periods, with simultaneous behavioral treatment administered for 60 minutes (additional 40 minutes following active tDCS).
  Interventions: Device: anodal right posterolateral cerebellar high-definition tDCS; Behavioral: computerized visual speech perception naming intervention
- Sham tDCS (Sham Comparator): For sham tDCS, electrodes were placed similarly, but the stimulator was turned off after a 30-second ramp-up and ramp-down period. Five session, similar procedures for the paired behavioral intervention.
  Interventions: Device: anodal right posterolateral cerebellar high-definition tDCS; Behavioral: computerized visual speech perception naming intervention

INTERVENTIONS:
Device: anodal right posterolateral cerebellar high-definition tDCS — Intervention delivered in two phases (active tDCS or sham tDCS first, order of treatment randomized across participants). Cerebellar tDCS: delivered using a Soterix Medical MxN High Definition tDCS Stimulator.
  Real tDCS applied to the right posterolateral cerebellum, with one anodal electrode (2 mA) placed at PO10 and two return electrodes (-1 mA each) at P10 and O10, using EEG-sized electrodes (external diameter of 1.2 cm) secured in an EEG cap. Participants received five sessions of tDCS combined with 60-min behavioral treatment. Real tDCS: delivered in the first 20 minutes of the behavioral intervention, 2 mA anodal stimulation with 30-second ramp-up and ramp-down periods.
  Sham tDCS - delivered using a Soterix Medical MxN High Definition tDCS Stimulator with similar montage as the active condition. Electrodes were placed similarly, but the stimulator was turned off after a 30-second ramp-up and ramp-down period.
Behavioral: computerized visual speech perception naming intervention — Computerized Naming Treatment: five consecutive 60-minute sessions. The computerized naming treatment adapted to Cantonese from Fridriksson et al. and delivered using DMDX. Lexical-semantic processing is engaged by providing auditory and visual articulatory cues. DMDX featured 100 Cantonese picture stimuli (50 objects and 50 actions), which have norms for timed-picture- naming in Cantonese. Participants viewed a black-and-white image of an item for 2 seconds, followed by a video showing the lower part of a speaker's face (nose and mouth) articulating the corresponding word. Participants then had up to 7 seconds to judge whether the picture stimulus matched the audio-visual presentation by pressing a "correct" or "incorrect" button.

SUMMARY:
The goal of this clinical trial is to learn if adding brain stimulation (cerebellar anodal tDCS) helps a computer-based therapy improve word-finding in Cantonese-speaking adults with aphasia after stroke. It will also check if the stimulation is safe and comfortable.

The main questions it aims to answer are:

Does real brain stimulation during therapy help people name pictures (both objects and actions) better and faster than fake (sham) stimulation?

Are there different effects on naming nouns (objects) versus verbs (actions)? Do any participants feel side effects like tingling or discomfort from the stimulation?

Researchers will compare real brain stimulation to sham (fake) stimulation while everyone gets the same 5-day computer therapy.

Participants will:

Do 60 minutes of computer word-naming practice every day for 5 days, twice (once with real stimulation, once with sham), with at least 2 weeks break in between

Wear a cap with electrodes on the back of the head for the first 20 minutes of each session to receive either real or sham brain stimulation

Name pictures on a computer before and after each 5-day block to measure improvement

Report any feelings or side effects after each session

DETAILED DESCRIPTION:
Aphasia is a frequent consequence of stroke, affecting about one-third of survivors and leading to significant emotional distress, functional limitations, and reduced social participation, all of which diminish quality of life. Speech-language therapy remains the primary treatment for language impairments, but its effectiveness varies considerably, and recovery is often incomplete. Non-invasive brain stimulation techniques, particularly transcranial direct current stimulation (tDCS), have emerged as promising adjuncts to therapy due to their portability, low cost, ease of use, and ability to enhance neural plasticity and cortical excitability in a polarity-dependent manner (anodal for excitation, cathodal for inhibition).

Traditionally, tDCS has targeted left-hemisphere cortical language areas, but post-stroke brain damage can disrupt current flow due to lesions and fluid accumulation. This has shifted attention to the cerebellum, which is often spared in aphasia, plays roles in linguistic and cognitive processing (especially right posterolateral regions), and connects to language networks. Despite its potential, few studies have examined cerebellar tDCS combined with language therapy for post-stroke aphasia, with existing evidence mostly from small trials in Western languages and limited data on tonal languages like Cantonese.

Additional Technical Information on the Methods

1. Study design: This study employs a randomized, double-blind, sham-controlled, crossover clinical trial design: participants randomly assigned to either the "tDCS-first" or "sham-first" group; both participants and researchers administering clinical testing and treatment blinded to the type of tDCS delivered until data analysis is concluded and, two independent study coordinators conduct the randomization and facilitate the setup for either active or sham tDCS sessions. Each treatment phase consists of five consecutive daily sessions, in which participants receive 60-minute-computerized naming treatment, with the first 20 minutes involving either active or sham tDCS. A 2-week washout period separates the two phases to minimize carryover effects.
2. Outcome measures:

   Timed confrontation naming task comprising 120 picture stimuli from the Object and Action Naming Battery (OANB) using the DMDX software for data collection. Each trial starts with a central fixation point displayed for 500 ms, followed immediately by a single picture stimulus presented centrally on the screen. The stimulus remains visible until a response is detected or 5000 ms had elapsed. DMDX records an error if no response is produced within the 2000 ms time limit. The task consisted of 60 trained and 60 untrained words, matched for imageability.
3. Computerized Naming Treatment - described in "Arms and Interventions" The 60-minute computerized naming treatment was adapted to Cantonese from Fridriksson et al. and delivered using DMDX. The treatment engages all domains of lexical-semantic processing by providing auditory and visual articulatory cues. The program features 100 Cantonese picture stimuli (50 objects and 50 actions) from the OANB, 60 of which included in the outcome naming task (trained items).
4. Adverse effects questionnaire: Participants were asked about adverse effects such as pain and/or discomfort (e.g., itching, irritation, tingling, or burning) before and after each session. The Wong-Baker FACES Pain Rating Scale was used to assess any tDCS-related discomfort.
5. tDCS protocol Cerebellar tDCS was delivered using a Soterix Medical MxN High Definition tDCS Stimulator. Intervention described in "Arms and Interventions"

Additional Technical Information on Data Analysis:

R version 4.4.1 used to the statistical analyses on the effects of intervention on naming accuracy and Reaction time (RT). Responses audio-recorded and reviewed for suitability prior to RT analysis; stimuli excluded from the RT analysis if contaminated by extraneous sounds before naming (e.g., coughs, starters, or fillers) or when the response provided is incorrect. RT outliers exceeding 3 standard deviations (SD) from the participants' means removed. Generalized linear mixed-effects models run to assess naming accuracy, while linear mixed-effects (LME) models utilized to evaluate naming RT for correct responses. T-tests employed to compare adverse effects between the sham and active conditions. Individual variability assessed by plotting performance for visual inspection of accuracy and mean RT raw scores and McNemar's test to evaluate changes in naming accuracy for each participant across time (pre- vs. immediate post-treatment), condition (active vs. sham), and grammatical category (nouns vs. verbs).

ELIGIBILITY:
Inclusion Criteria:

* Native Cantonese speakers
* Age: 40-80 years
* Diagnosed with aphasia
* Single left-hemispheric stroke ≥6 months prior
* Premorbid right-handedness
* Normal or corrected-to-normal vision
* Functional hearing (with or without hearing aids)

Exclusion Criteria:

* History of brain surgery
* Seizures within past 12 months
* Conditions contraindicated for tDCS (e.g., metallic implants, pacemakers)
* Prior neurological treatment (other than stroke-related)
* Severe cognitive impairment
* Naming accuracy <10% or >80% on noun/verb naming screening pretestt.

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2024-01-03 (Actual); Primary Completion 2024-04-15 (Actual); Study Completion 2025-06-01 (Actual)

PRIMARY OUTCOMES:
Accuracy on a timed confrontation naming task | - The baseline assessment on 'Day 1' - Outcome measure on 'Day 5'. - Data will be reported "through study completion, an average of 1 year"
  The timed confrontation naming task comprises 120 picture stimuli from the Object and Action Naming Battery (OANB) and is set for data collection using DMDX . Participants are instructed to name displayed pictures as quickly and ac-curately as possible using a microphone. Each trial started with a central fixation point displayed for 500 ms, followed immediately by a single picture stimulus presented centrally on the screen. The stimulus remains visible until a response is detected or 5000 ms have elapsed. DMDX records an error if no response was produced within the 2000 ms time limit.
  The naming task consists of 60 trained and 60 untrained words, half of them nouns and the other half verbs.
Reaction Time on a timed confrontation naming task | - The baseline assessment on 'Day 1' - Outcome measure on 'Day 5'. - Data will be reported "through study completion, an average of 1 year"
  The timed confrontation naming task comprises 120 picture stimuli from the Object and Action Naming Battery (OANB) and is set for data collection using DMDX . Participants are instructed to name displayed pictures as quickly and ac-curately as possible using a microphone. Each trial started with a central fixation point displayed for 500 ms, followed immediately by a single picture stimulus presented centrally on the screen. The stimulus remains visible until a response is detected or 5000 ms have elapsed. DMDX records an error if no response was produced within the 2000 ms time limit.
  The naming task consists of 60 trained and 60 untrained words, half of them nouns and the other half verbs.

CONTACTS AND LOCATIONS:
Overall Officials: Mehdi Bakhtiar, PhD, Principal Investigator — The University of Hong Kong
Locations (2):
- Hong Kong (2):
  - The University of Hong Kong, Hong Kong, Hong Kong SAR
  - Speech and Neuromodulation Lab, Hong Kong

IPD SHARING:
Plan to Share IPD: No